CLINICAL TRIAL: NCT04018690
Title: Project Arthritis Recovering Quality of Life Through Education - Hip
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, Full Professor in Orthopedics and Traumatology, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04019418700000068
Record Dates: First submitted 2019-06-27; First posted 2019-07-12 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis; Quality of Life; Function; Viscosuplementação
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — hylan; Ropivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): 24 patients with K&L 2 and 3 hip OA will be submitted to needle lavage, followed by the injection of 3mL of hylan, 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine.
  Interventions: Behavioral: Patients will be submitted to needle lavage, followed by the injection of 3mL of hylan and 1 mL of ropivacaine
- Control Group (Active Comparator): 24 patients with K&L 2 and 3 hip OA will be submitted to needle lavage, followed by the injection of 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine
  Interventions: Behavioral: Patients will be submitted to needle lavage, followed by the injection of 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine,

INTERVENTIONS:
Behavioral: Patients will be submitted to needle lavage, followed by the injection of 3mL of hylan and 1 mL of ropivacaine — Patients with K&L 2 and 3 hip OA will be submitted to needle lavage, followed by the injection of 3mL of hylan, 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine.
  Answer: WOMAC, Lequesne, VAS, EQ-5D-5L at inclusion, one week prior to surgery, 1st, 3rd, 6th and 12th months postoperatively.
  Submitted to evaluaton in the isokinetic dynamometer (Cybex 6000, Ronkokoma Lumex Inc.) where de amplitudes of movement of hip flexion, extension, abduction and adduction will be measures. Hip flexion, extension, abduction and adduction force will be assessed isokinetically at 60 degrees/second.
  Costs will be evaluated for cost-effectiveness and cost-utility analysis.
  Arms: Experimental
Behavioral: Patients will be submitted to needle lavage, followed by the injection of 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine, — Patients with K&L 2 and 3 hip OA will be submitted to needle lavage, followed by the injection of 0,5mL triamcinolone (10mg) and 1 mL of ropivacaine.
  Answer: WOMAC, Lequesne, VAS, EQ-5D-5L at inclusion, one week prior to surgery, 1st, 3rd, 6th and 12th months postoperatively.
  Submitted to evaluaton in the isokinetic dynamometer (Cybex 6000, Ronkokoma Lumex Inc.) where de amplitudes of movement of hip flexion, extension, abduction and adduction will be measures. Hip flexion, extension, abduction and adduction force will be assessed isokinetically at 60 degrees/second.
  Costs will be evaluated for cost-effectiveness and cost-utility analysis.
  Arms: Control Group

SUMMARY:
Introduction: One in four people are at risk of developing symptomatic hip OAH. Perhaps the greatest potential for improvement in OAH treatment is to approach the early stages of pathology, since total hip arthroplasty was considered 20th century surgery, with high cost-effectiveness in patients who are not responding to clinical treatment.

Joint lavage with saline shows significant pain relief in patients with knee and hip OA. In addition, when the saline solution is injected under pressure, it can generate a hydraulic distension of the capsule, increasing the joint amplitude and increasing the effect of drugs injected after washing. Injection of corticosteroids (CS) is recognized for improving the effects of joint washing, pain and even viscosupplementation.

In the investigators experience, lavage and infiltration of triamcinolone, lidocaine with or without hyaluronic acid led to subjective-functional improvement and range of motion of the majority of patients with OAH grades 2 and 3 of K & L undergoing the procedure. Intra-articular injection of hyaluronic acid (HA) is analgesic and anti-inflammatory in addition to promoting better distribution of forces, lowering pressure by weight and recovering the viscoelastic properties of synovial fluid, i.e., mechanical effects. In previous studies by the investigators, the addition of hilano to the lavage and injection of triamcinolone and local anesthetic led to gains in joint amplitude that were maintained over a year.

Objective: To evaluate whether lavage followed by injection of triamcinolone, ropivacaine and 4 mL of hylan in the affected joint (Hilano) improves function, range of motion, pain, quality of life and muscle strength in patients with OAH in the early stages METHODS: 48 patients from the public network attended by the Orthopedics and Traumatology Institute of the General Hospital of the Medical School of the University of São Paulo, already identified with bilateral OA of the hip submitted to THR in one limb and the other limb presenting OA mild or moderate with indication of non-surgical treatment will be submitted to lavage, saline infiltration and CS (control group) or lavage, saline infiltration, CS and Hilano. Patients will be assessed at 1, 3, 6 and 12 months after the procedure using standardized questionnaires (WOMAC and Lequesne), quality of life scales (Euroqol-EQ-5D-5L), pain, range of motion and strength using an isokinetic dynamometer.

DETAILED DESCRIPTION:
Hip OA (OAH) is less frequent than that of the hand and knee OA. One in four people have the risk of developing symptomatic OA of the hip.

Most guidelines for OAQ treatment combine recommendations for the treatment of knee and hip OA although OAH has specific etiopathogenic characteristics with its implications for individual therapeutic approaches.

Perhaps the greatest potential for improvement in OAH treatment is to approach the early stages of pathology, since total hip arthroplasty was considered to be 20th-century surgery with high cost-effectiveness in patients who are not responding to the clinical treatment of OA.

Measures that decrease inflammation and release capsular retraction leading to symptoms of pain and restriction of joint amplitude may improve the quality of life of these patients in the earliest stages of the disease.

Joint lavage with saline shows significant relief of pain in patients with knee and hip OA, probably by intra-articular removal of debris and factors that cause irritation and inflammation. In addition, when the saline solution is injected under pressure, it can generate a hydraulic distension of the capsule, increasing the joint amplitude and increasing the effect of drugs injected after washing. Injection of corticosteroids (CS) is recognized for improving the effects of joint washing, pain and even viscossuplementation.

In our experience, lavage and infiltration of triamcinolone, lidocaine with or without hyaluronic acid led to subjective-functional improvement and range of motion of most patients with OAH grades 2 and 3 of Kellgren and Lawrence undergoing the procedure.

The viscossuplementation of the hip has not yet been established in regard to type, dose, indication or frequency, and the number of existing jobs is relatively small in relation to those performed on knee osteoarthritis (OAK). Intra-articular injection of hyaluronic acid (HA) is analgesic and anti-inflammatory in addition to promoting better distribution of forces, lowering pressure by weight and recovering the viscoelastic properties of synovial fluid, i.e., mechanical effects. Its prolonged effect is explained by the action of hyaluronic acid on the CD44 receptors of synoviocytes and by the reduction of activated serum T cell levels. In our experience, the addition of hilano to the lavage and injection of triamcinolone and local anesthetic led to gains in joint amplitude that were maintained over a year.

Thus, the investigators developed a study to improve the range of motion and the function of patients with mild to moderate OA of the hip through lavage with physiological saline and hydraulic distension comparing to lavage, hydraulic distension and CS injection, anesthetic and a dose of 4mL of G-F20 hilano.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with bilateral OAH with or without comorbidities (metabolic syndrome, i.e. OA + at least two of overweight / central obesity, diabetes, dyslipidemia, hypertension)
* Age between 60 and 75 years who are awaiting primary THR, with indication of non-surgical treatment in the contralateral limb
* Patients without previous arthroplasties in the lower limbs.
* Patients with no personal history of chronic inflammatory arthritis (rheumatoid arthritis, for example).
* Patients with no personal history of cognitive, psychiatric and / or neurological disorders, whose symptoms presented at the time of evaluation are related or significantly interfere with the functions of attention, memory, logical reasoning, comprehension, in order to impair the assimilation of the given guidelines.
* Patients able to read, understand and respond to questionnaires and perform functional tests.

Exclusion Criteria:

* Fail to intervene and not perform the tasks determined by the professionals.
* Patients diagnosed during the study with chronic inflammatory arthritis (rheumatoid arthritis, for example)

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and ropivacaine improves range of flexion in the 3rd postoperative month in respect to lavage e triamcinolone injection. | 3 months
  Evaluate amplitudes of movement of hip flexion, extension, abduction and adduction; the hip flexion, extension, abduction and adduction force will be assessed isokinetically at 60 degrees / second.

SECONDARY OUTCOMES:
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine improves: Range of flexion, Range of motion (extension, adduction and abduction), Strength of flexion, extension, adduction e abduction. | 1 month, 6 months and 12 months
  Evaluate amplitudes of movement of hip flexion, extension, abduction and adduction; the hip flexion, extension, abduction and adduction force will be assessed isokinetically at 60 degrees / second.
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine improves: Womac | 1 month, 6 months and 12 months
  All patients will answer Womac questionnaire (Range minimum 0 - range maximum 96)
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine improves: Lequesne | 1 month, 6 months and 12 months
  All patients will answer Lequesne questionnaire (Range minimum 0 - range maximum 24)
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine improves: VAS | 1 month, 6 months and 12 months
  All patients will answer Visual Analogue Scale (Range minimum 0 - range maximum 100)
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine improves: EuroQol Questionnaire | 1 month, 6 months and 12 months
  All patients will answer EuroQol questionnaire
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine increases Lean Mass Percentage | 1 month, 6 months and 12 months
  Calculate lean mass of all patients
Evaluate whether needle lavage, followed by the injection of hylan, triamcinolone and 1 ropivacaine decrease fat percentage | 1 month, 6 months and 12 months
  Calculate fat percentage of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Ocampos, MD, Principal Investigator — University of São Paulo General Hospital
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813
- [Background] Murphy LB, Helmick CG, Schwartz TA, Renner JB, Tudor G, Koch GG, Dragomir AD, Kalsbeek WD, Luta G, Jordan JM. One in four people may develop symptomatic hip osteoarthritis in his or her lifetime. Osteoarthritis Cartilage. 2010 Nov;18(11):1372-9. doi: 10.1016/j.joca.2010.08.005. Epub 2010 Aug 14. PMID 20713163
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Rillo O, Riera H, Acosta C, Liendo V, Bolanos J, Monterola L, Nieto E, Arape R, Franco LM, Vera M, Papasidero S, Espinosa R, Esquivel JA, Souto R, Rossi C, Molina JF, Salas J, Ballesteros F, Radrigan F, Guibert M, Reyes G, Chico A, Camacho W, Urioste L, Garcia A, Iraheta I, Gutierrez CE, Aragon R, Duarte M, Gonzalez M, Castaneda O, Angulo J, Coimbra I, Munoz-Louis R, Saenz R, Vallejo C, Briceno J, Acuna RP, De Leon A, Reginato AM, Moller I, Caballero CV, Quintero M. PANLAR Consensus Recommendations for the Management in Osteoarthritis of Hand, Hip, and Knee. J Clin Rheumatol. 2016 Oct;22(7):345-54. doi: 10.1097/RHU.0000000000000449. PMID 27660931
- [Background] Murphy NJ, Eyles JP, Hunter DJ. Hip Osteoarthritis: Etiopathogenesis and Implications for Management. Adv Ther. 2016 Nov;33(11):1921-1946. doi: 10.1007/s12325-016-0409-3. Epub 2016 Sep 26. PMID 27671326
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Daigle ME, Weinstein AM, Katz JN, Losina E. The cost-effectiveness of total joint arthroplasty: a systematic review of published literature. Best Pract Res Clin Rheumatol. 2012 Oct;26(5):649-58. doi: 10.1016/j.berh.2012.07.013. PMID 23218429
- [Background] Chong T, Don DW, Kao MC, Wong D, Mitra R. The value of physical examination in the diagnosis of hip osteoarthritis. J Back Musculoskelet Rehabil. 2013;26(4):397-400. doi: 10.3233/BMR-130398. PMID 23948824
- [Background] de Sa D, Phillips M, Catapano M, Simunovic N, Belzile EL, Karlsson J, Ayeni OR. Adhesive capsulitis of the hip: a review addressing diagnosis, treatment and outcomes. J Hip Preserv Surg. 2015 Nov 27;3(1):43-55. doi: 10.1093/jhps/hnv075. eCollection 2016 Apr. PMID 27026818
- [Background] Ike RW, Arnold WJ, Rothschild EW, Shaw HL. Tidal irrigation versus conservative medical management in patients with osteoarthritis of the knee: a prospective randomized study. Tidal Irrigation Cooperating Group. J Rheumatol. 1992 May;19(5):772-9. PMID 1613709
- [Background] Chang RW, Falconer J, Stulberg SD, Arnold WJ, Manheim LM, Dyer AR. A randomized, controlled trial of arthroscopic surgery versus closed-needle joint lavage for patients with osteoarthritis of the knee. Arthritis Rheum. 1993 Mar;36(3):289-96. doi: 10.1002/art.1780360302. PMID 8452573
- [Background] Edelson R, Burks RT, Bloebaum RD. Short-term effects of knee washout for osteoarthritis. Am J Sports Med. 1995 May-Jun;23(3):345-9. doi: 10.1177/036354659502300317. PMID 7661265
- [Background] Vad VB, Sakalkale D, Warren RF. The role of capsular distention in adhesive capsulitis. Arch Phys Med Rehabil. 2003 Sep;84(9):1290-2. doi: 10.1016/s0003-9993(03)00261-2. PMID 13680563
- [Background] Vad VB, Sakalkale D, Sculco TP, Wickiewicz TL. Role of hylan G-F 20 in treatment of osteoarthritis of the hip joint. Arch Phys Med Rehabil. 2003 Aug;84(8):1224-6. doi: 10.1016/s0003-9993(03)00140-0. PMID 12917864
- [Background] Vad VB, Bhat AL, Sculco TP, Wickiewicz TL. Management of knee osteoarthritis: knee lavage combined with hylan versus hylan alone. Arch Phys Med Rehabil. 2003 May;84(5):634-7. doi: 10.1016/s0003-9993(02)04811-6. PMID 12736873
- [Background] Richette P, Ravaud P, Conrozier T, Euller-Ziegler L, Mazieres B, Maugars Y, Mulleman D, Clerson P, Chevalier X. Effect of hyaluronic acid in symptomatic hip osteoarthritis: a multicenter, randomized, placebo-controlled trial. Arthritis Rheum. 2009 Mar;60(3):824-30. doi: 10.1002/art.24301. PMID 19248105
- [Background] Ozturk C, Atamaz F, Hepguler S, Argin M, Arkun R. The safety and efficacy of intraarticular hyaluronan with/without corticosteroid in knee osteoarthritis: 1-year, single-blind, randomized study. Rheumatol Int. 2006 Feb;26(4):314-9. doi: 10.1007/s00296-005-0584-z. Epub 2005 Feb 10. PMID 15703953
- [Background] van Middelkoop M, Arden NK, Atchia I, Birrell F, Chao J, Rezende MU, Lambert RG, Ravaud P, Bijlsma JW, Doherty M, Dziedzic KS, Lohmander LS, McAlindon TE, Zhang W, Bierma-Zeinstra SM. The OA Trial Bank: meta-analysis of individual patient data from knee and hip osteoarthritis trials show that patients with severe pain exhibit greater benefit from intra-articular glucocorticoids. Osteoarthritis Cartilage. 2016 Jul;24(7):1143-52. doi: 10.1016/j.joca.2016.01.983. Epub 2016 Feb 2. PMID 26836288
- [Background] de Campos GC, Rezende MU, Pailo AF, Frucchi R, Camargo OP. Adding triamcinolone improves viscosupplementation: a randomized clinical trial. Clin Orthop Relat Res. 2013 Feb;471(2):613-20. doi: 10.1007/s11999-012-2659-y. Epub 2012 Oct 26. PMID 23100188
- [Background] Zhang W, Doherty M, Arden N, Bannwarth B, Bijlsma J, Gunther KP, Hauselmann HJ, Herrero-Beaumont G, Jordan K, Kaklamanis P, Leeb B, Lequesne M, Lohmander S, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Swoboda B, Varatojo R, Verbruggen G, Zimmermann-Gorska I, Dougados M; EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). EULAR evidence based recommendations for the management of hip osteoarthritis: report of a task force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2005 May;64(5):669-81. doi: 10.1136/ard.2004.028886. Epub 2004 Oct 7. PMID 15471891
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Gomis A, Pawlak M, Balazs EA, Schmidt RF, Belmonte C. Effects of different molecular weight elastoviscous hyaluronan solutions on articular nociceptive afferents. Arthritis Rheum. 2004 Jan;50(1):314-26. doi: 10.1002/art.11421. PMID 14730630
- [Background] Bagga H, Burkhardt D, Sambrook P, March L. Longterm effects of intraarticular hyaluronan on synovial fluid in osteoarthritis of the knee. J Rheumatol. 2006 May;33(5):946-50. PMID 16652425
- [Background] Gomis A, Miralles A, Schmidt RF, Belmonte C. Intra-articular injections of hyaluronan solutions of different elastoviscosity reduce nociceptive nerve activity in a model of osteoarthritic knee joint of the guinea pig. Osteoarthritis Cartilage. 2009 Jun;17(6):798-804. doi: 10.1016/j.joca.2008.11.013. Epub 2008 Nov 27. PMID 19103502
- [Background] Waddell DD, Kolomytkin OV, Dunn S, Marino AA. Hyaluronan suppresses IL-1beta-induced metalloproteinase activity from synovial tissue. Clin Orthop Relat Res. 2007 Dec;465:241-8. doi: 10.1097/BLO.0b013e31815873f9. PMID 18090474
- [Background] Balaz EA. Chemistry and biology of hyaluronan. In: Garg HG, Hales CA, editors. Chemistry and biology of hyaluronan. Elsevier; 2004. p. 415-55
- [Background] Wang CT, Lin YT, Chiang BL, Lin YH, Hou SM. High molecular weight hyaluronic acid down-regulates the gene expression of osteoarthritis-associated cytokines and enzymes in fibroblast-like synoviocytes from patients with early osteoarthritis. Osteoarthritis Cartilage. 2006 Dec;14(12):1237-47. doi: 10.1016/j.joca.2006.05.009. Epub 2006 Jun 30. PMID 16806998
- [Background] Julovi SM, Yasuda T, Shimizu M, Hiramitsu T, Nakamura T. Inhibition of interleukin-1beta-stimulated production of matrix metalloproteinases by hyaluronan via CD44 in human articular cartilage. Arthritis Rheum. 2004 Feb;50(2):516-25. doi: 10.1002/art.20004. PMID 14872494
- [Background] Yasuda T. Hyaluronan inhibits prostaglandin E2 production via CD44 in U937 human macrophages. Tohoku J Exp Med. 2010 Mar;220(3):229-35. doi: 10.1620/tjem.220.229. PMID 20208419
- [Background] Liu CC, Su LJ, Tsai WY, Sun HL, Lee HC, Wong CS. Hylan G-F 20 attenuates posttraumatic osteoarthritis progression: Association with upregulated expression of the circardian gene NPAS2. Life Sci. 2015 Nov 15;141:20-4. doi: 10.1016/j.lfs.2015.09.007. Epub 2015 Sep 24. PMID 26388558
- [Background] Lurati A, Laria A, Mazzocchi D, Re KA, Marrazza M, Scarpellini M. Effects of hyaluronic acid (HA) viscosupplementation on peripheral Th cells in knee and hip osteoarthritis. Osteoarthritis Cartilage. 2015 Jan;23(1):88-93. doi: 10.1016/j.joca.2014.09.010. Epub 2014 Sep 22. PMID 25246074
- [Background] Cliborne AV, Wainner RS, Rhon DI, Judd CD, Fee TT, Matekel RL, Whitman JM. Clinical hip tests and a functional squat test in patients with knee osteoarthritis: reliability, prevalence of positive test findings, and short-term response to hip mobilization. J Orthop Sports Phys Ther. 2004 Nov;34(11):676-85. doi: 10.2519/jospt.2004.34.11.676. PMID 15609488
- [Background] Singh J, Khan WS, Marwah S, Wells G, Tannous DK, Sharma HK. Do we need radiological guidance for intra-articular hip injections? Open Orthop J. 2014 May 16;8:114-7. doi: 10.2174/1874325001408010114. eCollection 2014. PMID 24893653
- [Background] Byrd JW. Hip arthroscopy utilizing the supine position. Arthroscopy. 1994 Jun;10(3):275-80. doi: 10.1016/s0749-8063(05)80111-2. PMID 8086020
- [Background] Byrd JW, Pappas JN, Pedley MJ. Hip arthroscopy: an anatomic study of portal placement and relationship to the extra-articular structures. Arthroscopy. 1995 Aug;11(4):418-23. doi: 10.1016/0749-8063(95)90193-0. PMID 7575873
- [Background] Schmidt-Braekling T, Waldstein W, Renner L, Valle AG, Bou Monsef J, Boettner F. Ultrasound and fluoroscopy are unnecessary for injections into the arthritic hip. Int Orthop. 2015 Aug;39(8):1495-7. doi: 10.1007/s00264-014-2648-8. Epub 2015 Jan 16. PMID 25592829